CLINICAL TRIAL: NCT06670508
Title: The Efficacy of Erector Spinae Block Versus Transversus Abdominis Plane Block in Laparoscopic Nephrectomy: Randomized Comparative Trial
Brief Title: The Efficacy of Erector Spinae Block Versus Transversus Abdominis Plane Block in Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Youssef Ollaek, Assisstant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS-95-2023
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Pain Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Active Comparator): Group A, The patient was in the supine position then; the TAP block was given by a high frequency linear ultrasound transducer (Siemens acuson x300 3-5MHz ultrasound). After skin preparation and isolation, the transducer was placed 2 cm sub-xiphoid, then moved along the subcostal edge to identify the rectus abdominis muscle and the transversus abdominis then, a blunted tip, 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) was introduced in-plane 2-3 cm lateral to the transducer, under direct ultrasound visualization. After confirming the correct placement of the needle and the negative aspiration probe, the rest of the anaesthetic substance was injected along the subcostal line in the transversus abdominis plane 20 ml 0.25% bupivacaine on each side after aspiration to avoid intravascular placement, and the dissection of the plane was observed. The block was performed bilaterally.
  Interventions: Procedure: Transversus Abdominis Plane block
- ES Block (Active Comparator): Group B, the patient was placed in the prone position. Then, the Erector Spinae block was given by same ultrasound transducer . It was sagittaly placed against the target vertebral level (T7 transverse process) in the prone position and moved in approximately 3-cm lateral to the spinous process.. The Erector Spinae muscle and transverse process was identified, and a same blunted tip , 20-gauge, short bevel needle was advanced, using the in-plane approach, in cephalad-to-caudal direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane. The block was performed bilaterally by injecting 40 mL of 0.25% bupivacaine (20 mL into each side) into the fascial plane between the deep surface of the Erector Spinae muscle and the transverse processes of the lumbar vertebrae laterally.
  Interventions: Procedure: Erector Spinae Plane block

INTERVENTIONS:
Procedure: Transversus Abdominis Plane block — Group A, The patient was in the supine position then; the TAP block was given by a high frequency linear ultrasound transducer (Siemens acuson x300 3-5MHz ultrasound). After skin preparation and isolation, the transducer was placed 2 cm sub-xiphoid, then moved along the subcostal edge to identify the rectus abdominis muscle and the transversus abdominis then, a blunted tip, 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) was introduced in-plane 2-3 cm lateral to the transducer, under direct ultrasound visualization. After confirming the correct placement of the needle and the negative aspiration probe, the rest of the anaesthetic substance was injected along the subcostal line in the transversus abdominis plane 20 ml 0.25% bupivacaine on each side after aspiration to avoid intravascular placement, and the dissection of the plane was observed. The block was performed bilaterally.
  Arms: TAP Block
Procedure: Erector Spinae Plane block — Group B, the patient was placed in the prone position. Then, the Erector Spinae block was given by same ultrasound transducer . It was sagittaly placed against the target vertebral level (T7 transverse process) in the prone position and moved in approximately 3-cm lateral to the spinous process.. The Erector Spinae muscle and transverse process was identified, and a same blunted tip , 20-gauge, short bevel needle was advanced, using the in-plane approach, in cephalad-to-caudal direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane. The block was performed bilaterally by injecting 40 mL of 0.25% bupivacaine (20 mL into each side) into the fascial plane between the deep surface of the Erector Spinae muscle and the transverse processes of the lumbar vertebrae laterally.
  Arms: ES Block

SUMMARY:
The investigators hypothesis that erector spinae block better than transversus abdominus plane block regarding the post operative pain management.

DETAILED DESCRIPTION:
Aim of the work:

The purpose of this study to compare erector spinae block to transversus abdominus plane block in laparoscopic nephrectomy regarding analgesic efficacy and postoperative morphine consumption.

Statistical Analysis

I. Sample size:

Sample size was calculated using G-power software. A previous study (reference) reported that the amount of morphine used in the first 6 hours in patients received TAP block in nephrectomy was 12.4 ± 8.4. Assuming that the amount will change by 50% at least with the other block, a power of 80% and an alpha error of 0.5, the minimum sample size required will be 60 patients (30 in each group). We will increase it to 35 in each group to compensate for drop-outs. (15)

II. Statistical analysis:

All measurement indexes will be expressed as mean ± SD/standard error of the mean or number (%). After analysis of normality of data distribution, normally distributed data will be compared by the independent sample t-test. Unpaired quantitative variables will be evaluated by the Student t-test and analysis of variance. The Mann-Whitney U test will be employed for intergroup comparison, and the Wilcoxon signed-rank test for comparison between different time points within the same group. Intergroup comparison of categorical variables will be performed by the chi-square test. Values of A P value less than 0.05 will be considered statistically significant. All data will be statistically analyzed by statisticians using the SPSS 16.0 software package (IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patient age (>18 and <60)
* Both sexes
* American Society of Anesthesiologists (ASA) physical status classes I and II
* Patients scheduled for laparoscopic nephrectomy surgery.

Exclusion Criteria:

* Refusal of regional block
* Patients with uncontrolled diabetes or hypertension
* Patients with neurological, psychological disorders or those lacking cooperation
* Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
* Patients with bleeding disorders defined as (INR >2) and/ or (platelet count <100,000/µL)
* Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
* Patients who are allergic to amide local anesthetics.
* Cases converted to open surgery will also be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The amount of morphine consumed within 6 hours postoperatively | Immediatly post operative for 6 hours
  The amount of morphine consumed within 6 hours postoperatively

SECONDARY OUTCOMES:
Failure rate in both groups | in first hour postoperatively
  Failure rate in both groups
Time taken to perform a successful block | 30 minutes from time just after local anesthetic injection to successful site of incisions and dermatomal coverage
  Time taken to perform a successful block
Postoperative nausea and vomiting | Immediatly post operative for 24 hours
  Incidence of postoperative nausea and vomiting
Time to ambulate in both groups | Immediate 24 hours post-operative
  Time to ambulate in both groups
p/f ratio postoperatively in both groups | after first 12, 24 hours postoperatively
  p/f ratio postoperatively in both groups
Incidence of postoperative pulmonary complication | chest x-ray Immediate 24 hours post-operative
  Incidence of postoperative pulmonary complication
Incidence of complications (hematoma at the site of injection and local anesthetic toxicity) related to each block | Immediate 24 hours post-operative
  Incidence of complications (hematoma at the site of injection and local anesthetic toxicity) related to each block
Time for first rescue analgesia in each block | Immediate 24 hours post-operative
  Time for first rescue analgesia in each block
Total opioid consumption in each block | Immediate 24 hours post-operative
  Total opioid consumption in each block

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ollaek, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Cairo, Egypt